CLINICAL TRIAL: NCT00005564
Title: Impact of Adult Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5113; R01HL056438 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To assess the separate and interactive effects of asthma severity, subspecialty practice variation, asthma-related psychosocial variables, and other factors on asthma outcomes, including asthma-specific quality of life and activity limitations, health care utilization for asthma, and direct and indirect costs of asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is both common and costly. Neither the risk factors of poor outcome nor the predictors of better outcome are well understood. Illness severity is clearly an important predictive factor in asthma, but may explain less variability in outcome than other determinants, such as patient-perceived asthma control, other asthma-related psychosocial measures, and the kind and extent of subspecialty care for asthma. By quantifying predictors of asthma-specific quality of life, functional status, services utilization, and the direct and indirect illness costs of asthma, this study addressed a major research gap in secondary and tertiary prevention efforts.

DESIGN NARRATIVE:

A random sample of pulmonary and allergy subspecialists initially enrolled 600 persons with asthma identified in patient visit logs. This established panel completed 45 minute baseline and follow-up computer-assisted telephone interviews (CATI); 539 (90%) were successfully re-interviewed after 18 months of follow-up. A supplemental sampling frame of persons with asthma identified from family practitioners was completed as was a group with rhinitis but without asthma. Interviews assessed disease severity and other covariables using validated survey instruments. Pulmonary function and medical records were used to validate severity in a sub-sample of subjects. The study extended longitudinal follow-up study of this initial cohort. Its analysis tested predictive models for the asthma outcomes of interest.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Blanc — University of California at San Francisco

REFERENCES:
- [Background] Katz PP, Eisner MD, Henke J, Shiboski S, Yelin EH, Blanc PD. The Marks Asthma Quality of Life Questionnaire: further validation and examination of responsiveness to change. J Clin Epidemiol. 1999 Jul;52(7):667-75. doi: 10.1016/s0895-4356(99)00026-8. PMID 10391660
- [Background] Yelin E, Henke J, Katz PP, Eisner MD, Blanc PD. Work dynamics of adults with asthma. Am J Ind Med. 1999 May;35(5):472-80. doi: 10.1002/(sici)1097-0274(199905)35:53.0.co;2-s. PMID 10212700
- [Background] Eisner MD, Katz PP, Yelin EH, Henke J, Smith S, Blanc PD. Assessment of asthma severity in adults with asthma treated by family practitioners, allergists, and pulmonologists. Med Care. 1998 Nov;36(11):1567-77. doi: 10.1097/00005650-199811000-00006. PMID 9821944
- [Background] Eisner MD, Yelin EH, Henke J, Shiboski SC, Blanc PD. Environmental tobacco smoke and adult asthma. The impact of changing exposure status on health outcomes. Am J Respir Crit Care Med. 1998 Jul;158(1):170-5. doi: 10.1164/ajrccm.158.1.9801028. PMID 9655725 (Retraction: PMID 10988082 Eisner MD, Shiboski SC, Yelin EH, Blanc PD, Bainton DF. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):788)
- [Background] Eisner MD, Yelin EH, Katz PP, Shiboski SC, Henke J, Blanc PD. Predictors of cigarette smoking and smoking cessation among adults with asthma. Am J Public Health. 2000 Aug;90(8):1307-11. doi: 10.2105/ajph.90.8.1307. PMID 10937016
- [Background] Yelin E, Trupin L, Cisternas M, Eisner M, Katz P, Blanc P. A national study of medical care expenditures for respiratory conditions. Eur Respir J. 2002 Mar;19(3):414-21. doi: 10.1183/09031936.02.00522001. PMID 11936516
- [Background] Blanc PD, Trupin L, Earnest G, Katz PP, Yelin EH, Eisner MD. Alternative therapies among adults with a reported diagnosis of asthma or rhinosinusitis : data from a population-based survey. Chest. 2001 Nov;120(5):1461-7. doi: 10.1378/chest.120.5.1461. PMID 11713120
- [Background] Eisner MD, Katz PP, Yelin EH, Shiboski SC, Blanc PD. Risk factors for hospitalization among adults with asthma: the influence of sociodemographic factors and asthma severity. Respir Res. 2001;2(1):53-60. doi: 10.1186/rr37. Epub 2000 Dec 29. PMID 11686864
- [Background] Eisner MD, Katz PP, Yelin EH, Hammond SK, Blanc PD. Measurement of environmental tobacco smoke exposure among adults with asthma. Environ Health Perspect. 2001 Aug;109(8):809-14. doi: 10.1289/ehp.01109809. PMID 11564616
- [Background] Blanc PD, Trupin L, Eisner M, Earnest G, Katz PP, Israel L, Yelin EH. The work impact of asthma and rhinitis: findings from a population-based survey. J Clin Epidemiol. 2001 Jun;54(6):610-8. doi: 10.1016/s0895-4356(00)00349-8. PMID 11377122
- [Background] Katz PP, Yelin EH, Eisner MD, Blanc PD. Perceived control of asthma and quality of life among adults with asthma. Ann Allergy Asthma Immunol. 2002 Sep;89(3):251-8. doi: 10.1016/S1081-1206(10)61951-5. PMID 12269644
- [Background] Eisner MD, Yelin EH, Katz PP, Earnest G, Blanc PD. Exposure to indoor combustion and adult asthma outcomes: environmental tobacco smoke, gas stoves, and woodsmoke. Thorax. 2002 Nov;57(11):973-8. doi: 10.1136/thorax.57.11.973. PMID 12403881
- [Background] Eisner MD, Blanc PD. Environmental tobacco smoke exposure during travel among adults with asthma. Chest. 2002 Sep;122(3):826-8. doi: 10.1378/chest.122.3.826. PMID 12226020
- [Background] Blanc PD, Trupin L, Earnest G, San Pedro M, Katz PP, Yelin EH, Eisner MD. Effects of physician-related factors on adult asthma care, health status, and quality of life. Am J Med. 2003 May;114(7):581-7. doi: 10.1016/s0002-9343(03)00053-6. PMID 12753882
- [Background] Cisternas MG, Blanc PD, Yen IH, Katz PP, Earnest G, Eisner MD, Shiboski S, Yelin EH. A comprehensive study of the direct and indirect costs of adult asthma. J Allergy Clin Immunol. 2003 Jun;111(6):1212-8. doi: 10.1067/mai.2003.1449. PMID 12789219
- [Background] Snyder L, Blanc PD, Katz PP, Yelin EH, Eisner MD. Leukotriene modifier use and asthma severity: how is a new medication being used by adults with asthma? Arch Intern Med. 2004 Mar 22;164(6):617-22. doi: 10.1001/archinte.164.6.617. PMID 15037489